CLINICAL TRIAL: NCT01023711
Title: Assessment of the Effect of Age and Priming on the Immunological Response to an Inactivated Vaccine for Novel H1N1 Virus.
Brief Title: Immunologic Response to Inactivated Vaccine for Novel H1N1 Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, John Treanor, MD, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URMC 09-005
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inactivated H1N1 Vaccine (Other): Subject will recieve 0.5 mL IM injection of Inactivated H1N1 vaccine
  Interventions: Biological: Inactivated H1N1 vaccine

INTERVENTIONS:
Biological: Inactivated H1N1 vaccine — 0.5 ml IM into Deltoid region of arm
  Other Names: Influenza A (H1 N1) 2009 Monovalent Vaccine
Biological: Inactivated H1N1 vaccine — 0.5 mL IM X 1 dose
  Other Names: Swine Flu Vaccine

SUMMARY:
The purpose of this study is to describe the immune response to a novel H1N1 influenza vaccination in healthy adults, and to understand the factors that allow healthy adults to respond to a single dose of vaccine even if they have never previously experience novel H1N1 disease or vaccination.

DETAILED DESCRIPTION:
Studies have now determined that only a single dose of inactivated vaccine is needed for immunization against novel H1N1, but the reasons why adults appear to be ready to respond to a single dose are not known.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-32 years, or 60 years and older
* No history of Novel H1N1 virus or vaccine
* Female not able to bear children or not pregnant and agrees to practice effective birth control
* Female negative pregnancy test
* Good Health
* Ability to understand and comply with protocol
* Provided Informed Consent

Exclusion Criteria:

* Previous history of vaccination against novel H1N1 or laboratory documented H1N1 infection
* Previous history of vaccination with A/New Jersey/76 vaccine (for subjects 60 & older
* History of egg allergy or is allergic to other components of the vaccine
* Women who are pregnant or breastfeeding or intends to get pregnant during the study period between enrollment & 30 days following vaccination
* Subject is immunosuppressed as the result of underlying illness or treatment with immunosuppressive or cytotoxic drugs or use of chemotherapy/radiation therapy in the preceding 36 months
* Subject has active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy. "Active" is defined as treatment within the past 5 years.
* Long term (greater than 2 weeks) use of oral or parental steroids, or high- dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal & topical steroids allowed)
* Received immunoglobulin or other blood product within 3 months prior to enrollment in this study
* Subject has received an inactivated vaccine within 2 weeks or a live vaccine within 4 weeks prior to enrollment or plans to receive another vaccine within the next 28 days
* Subject has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. Those conditions include chronic conditions recognized as risk factors for influenza complications or as contraindicated for live vaccination, including chronic cardiac (exclusive of hypertension) or pulmonary conditions (including asthma), diabetes mellitus, or renal impairment
* Subject has an acute illness or an oral temperature greater then 99.9 F(37.7 C)within 3 days of enrollment or vaccination. Subject who has acute illness that was treated, symptoms resolved are eligible to enroll as long as treatment is complete & symptoms resolved > 3 days prior to enrollment.
* Subject is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month of enrollment in this study, or intends to donate blood during this period.
* Subject has any condition that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
* Subject has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis, or are receiving psychiatric drugs. Subjects who are receiving a single anti-depressant drug & are stable for at least 3 months prior to enrollment without decompensation are allowed enrollment into the study.
* Subject has a history of alcohol or drug abuse in the 5 years of enrollment.
* Subject has known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Subject has a previous history of Guillain-Barre syndrome within 6 weeks of receipt of influenza vaccine
* Subject has any condition that the principal investigator (PI) believes may interfere with the successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Treanor, M.D., Principal Investigator — University of Rochester
Locations (1):
- Vaccine Research Unit Room 3-5000, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via flyers and advertisments. Recruitment began 12/2009 and ended 10/2010. Subjects were screened via IRB approved Screening script by phone and visit as indicated.
Pre-assignment Details: Subjects 18-32 were required to have a serum antibody test done during screening. Their HAI antibody level needed to be less than or = to 1:8. Female subjects of childbearing potential must have a negative pregnancy test at screening.
Groups:
- H1N1 Monovalent Influenza Vaccine: 0.5 mL IM of Influenza A (H1N1) 2009 Monovalent Vaccine
Period: Overall Study
Arm/Group | H1N1 Monovalent Influenza Vaccine
Started | 107
Completed | 107
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | H1N1 Monovalent Influenza Vaccine
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.19626 (21.47638)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Determination of Immune Response to Vaccination.
Description: Number of participants with a 4-fold or greater increase in serum HAI antibody from pre- to 28 day post-vaccination
Time Frame: 28 days
Population: All subjects who completed Day 28 visit post vaccination were analyzed.
Measure: Number; unit: participants
Arm/Group | H1N1 Monovalent Influenza Vaccine
Number analyzed (Participants) | 55
participants | 45

2. Secondary Outcome: Assessment of the Reactogenicity Events Post Vaccination.
Description: Number of subjects with reactogenicity events of grade 2 or higher within 7 days of vaccination
Time Frame: 7 days
Population: Subjects who completed the 7 day diary card
Measure: Number; unit: participants
Arm/Group | Inactivated H1N1 Vaccine
Number analyzed (Participants) | 58
participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events both non-serious and serious were collected from Day O (day of vaccination thru day 28. Reactogenicity events were collected on a memory aid from day 0 to day 7.
Arm/Group | H1N1 Monovalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 14/107
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H1N1 Monovalent Influenza Vaccine (N=107)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 8 (8)
FATIGUE (General disorders) | 3 (3)
CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No